CLINICAL TRIAL: NCT03265327
Title: The Use of a Novel Oral Supplement Containing Omega-3 and Omega-6 Fatty Acids on Dry Eye Symptoms (TURMERIC)
Brief Title: Effect of an Oral Supplement Containing Omega-3 and Omega-6 on Dry Eye Symptoms
Acronym: TURMERIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nature's Way Canada (Industry)
Collaborators: Centre for Contact Lens Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22309
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Subjects will receive an oral supplement containing fish oil, evening primrose oil and borage oil.
  Interventions: Dietary Supplement: Oral supplement containing omega-3 and omega-6
- Placebo (Placebo Comparator): Subjects will receive an oral supplement containing coconut oil and light olive oil.
  Interventions: Dietary Supplement: Oral supplement containing coconut and olive oil

INTERVENTIONS:
Dietary Supplement: Oral supplement containing omega-3 and omega-6 — An oral supplement containing omega-3 and omega-6
  Arms: Treatment
Dietary Supplement: Oral supplement containing coconut and olive oil — An oral supplement containing coconut oil and olive oil
  Arms: Placebo

SUMMARY:
This study will investigate the effectiveness of two oral supplements on the ocular signs and symptoms in symptomatic dry eye patients. Eligible participants will be given one of two oral supplements to take once a day for up to three months.

ELIGIBILITY:
Inclusion Criteria:

1. Is over 19 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and anticipated to be able to comply with the daily intake of liquid oil supplements (one teaspoon per day for three months);
4. Is willing and able to follow instructions and maintain the appointment schedule;
5. Exhibit moderate ocular dryness symptoms, defined as:

   1. A score of ≥23 on the Ocular Surface Disease Index (OSDI, (Allergan Inc., Irvine, CA)) questionnaire;
   2. Currently uses, or feels the need to use eye drops to relieve symptoms of dryness.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Currently wears, or has worn contact lenses in the past 3 months;
4. Has sensitivity or an allergy to products that contain fish, soy, coconut oil or olive oil;
5. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
6. Is using any systemic or topical medications (including topical corticosteroids/NSAIDs or glaucoma medications) that in the opinion of the investigator may affect a study outcome variable;
7. Is currently taking, or has used, any omega-3 or omega-6 supplements in the last three months;
8. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
9. Is pregnant, lactating or planning a pregnancy at the time of enrolment;
10. Is aphakic;
11. Has undergone refractive error surgery;
12. Is an employee of the Centre for Contact Lens Research;
13. Has taken part in another (pharmaceutical) research study within the last 30 days;

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) score | At screening
  The OSDI is assessed on a scale of 0 and 100. A higher composite score indicates more severe dryness.
Ocular Surface Disease Index (OSDI) score | At 1 month
  The OSDI is assessed on a scale of 0 and 100. A higher composite score indicates more severe dryness.
Ocular Surface Disease Index (OSDI) score | At 3 months
  The OSDI is assessed on a scale of 0 and 100. A higher composite score indicates more severe dryness.
Symptom Assessment in Dry Eye (SANDE) questionnaire | At screening
  The Symptom Assessment in Dry Eye (SANDE) questionnaire is a dry eye questionnaire that asks participants to describe the frequency and severity of their dry eye symptoms using a visual analogue scale.
Symptom Assessment in Dry Eye (SANDE) questionnaire | At 1 month
  The Symptom Assessment in Dry Eye (SANDE) questionnaire is a dry eye questionnaire that asks participants to describe the frequency and severity of their dry eye symptoms using a visual analogue scale.
Symptom Assessment in Dry Eye (SANDE) questionnaire | At 3 months
  The Symptom Assessment in Dry Eye (SANDE) questionnaire is a dry eye questionnaire that asks participants to describe the frequency and severity of their dry eye symptoms using a visual analogue scale.
Schirmers test | At screening
  The small strip of paper is removed from the Schirmer test package, folded at one end, and is inserted into the outer corner of the participant's eyes. The participant is asked to close their eyes and wait for 5 minutes. After 5 minutes, the paper is removed and the length of which the paper strip is wetted is recorded in mm.
Schirmers test | At 1 month
  The small strip of paper is removed from the Schirmer test package, folded at one end, and is inserted into the outer corner of the participant's eyes. The participant is asked to close their eyes and wait for 5 minutes. After 5 minutes, the paper is removed and the length of which the paper strip is wetted is recorded in mm.
Schirmers test | At 3 months
  The small strip of paper is removed from the Schirmer test package, folded at one end, and is inserted into the outer corner of the participant's eyes. The participant is asked to close their eyes and wait for 5 minutes. After 5 minutes, the paper is removed and the length of which the paper strip is wetted is recorded in mm.
Objective non-invasive tear film stability (NIKBUT) | At screening
  Time taken for tear film breakup as measured objectively in seconds.
Objective non-invasive tear film stability (NIKBUT) | At 1 month
  Time taken for tear film breakup as measured objectively in seconds.
Objective non-invasive tear film stability (NIKBUT) | At 3 months
  Time taken for tear film breakup as measured objectively in seconds.
Non-invasive tear break up time (NITBUT) | At screening
  Time taken for tear film breakup as measured by a study investigator in seconds.
Non-invasive tear break up time (NITBUT) | At 1 month
  Time taken for tear film breakup as measured by a study investigator in seconds.
Non-invasive tear break up time (NITBUT) | At 3 months
  Time taken for tear film breakup as measured by a study investigator in seconds.

SECONDARY OUTCOMES:
Change in Bulbar hyperemia after 3 months | At screening, 1 month and 3 months
  The redness of the bulbar conjunctiva of both eyes will be assessed in all four quadrants using the Efron scale (0-4, in 0.1 steps).
Change in Limbal hyperemia after 3 months | At screening, 1 month and 3 months
  The redness of the limbal conjunctiva of both eyes will be assessed in all four quadrants using the Efron scale (0-4, in 0.1 steps).
Change in Tear meniscus height after 3 months | At screening, 1 month and 3 months
  Measurement of tear meniscus height in mm.
Change in Meiboscore (Arita's scale) after 3 months | At screening, 1 month and 3 months
  Graded on 0-3 scale. Grade 0: no dropout, Grade 1: < 1/3 total area dropout, Grade 2: 1/3 to 2/3 total area dropout, Grade 3: > 2/3 total area dropout
Change in Visual acuity after 3 months | At screening, 1 month and 3 months
  High contrast logMAR VA with computerized charts in high illumination
Change in Tear osmolarity after 3 months | At screening and 3 months
  Measure of the osmolarity of collected tears.
Change in Omega-3 index after 3 months | At screening and 3 months
  Amount of EPA and DHA in erythrocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng A, Woods J, Jahn T, Jones LW, Sullivan Ritter J. Effect of a Novel Omega-3 and Omega-6 Fatty Acid Supplement on Dry Eye Disease: A 3-month Randomized Controlled Trial. Optom Vis Sci. 2022 Jan 1;99(1):67-75. doi: 10.1097/OPX.0000000000001826. PMID 34882608